CLINICAL TRIAL: NCT00759486
Title: Pediatric Facial Fracture Growth and Development Study
Brief Title: Pediatric Facial Fracture Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Joseph Losee, Ross H. Musgrave Professor of Pediatric Plastic Surgery Executive Vice-Chair and Program Director Department of Plastic Surgery University of Pittsburgh Medical Center, University of Pittsburgh
Other Study IDs: 0509046
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Craniofacial Fracture
Keywords: craniofacial fracture; Subjects who are in the active phase of craniofacial skeletal growth, and have sustained a craniofacial fracture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is to establish a prospective, long-term, comprehensive growth and development study of the pediatric craniofacial skeleton following fracture, whose recruitment is ongoing.

DETAILED DESCRIPTION:
This is a prospective, long-term, comprehensive growth and development study of the pediatric craniofacial skeleton following fracture.

This study will encompass two specific aims:

1. To compare the growth and development of the pediatric craniofacial skeleton after fracture to publish standardized means of dentofacial growth in the Bolton-Brush Growth Study. Patients will be matched according to age, gender, and ethnicity. The status of dental eruption will be recorded as well as the vertical and anteroposterior classification of occlusion. The effect of trauma on the eruption and vitality of permanent teeth will be recorded. We will further assess the popularly held theories of craniofacial growth and effects of injury to various facial growth sites (i.e. mandibular condyles, nasal septum).
2. Attempt to evaluate the effects of various treatment modalities of facial fracture on skeletal growth and development (i.e. open reduction and internal fixation versus closed reduction and external fixation), (open reduction and internal fixation with metallic vs. absorbable fixation). We will evaluate the effect of metallic internal fixation on subsequent craniofacial skeletal growth and development, as well as the routine needed for its removal.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion in the research study will be any pediatric patient, birth to 18 years, who are in the active phase of craniofacial skeletal growth, and have sustained a craniofacial fracture.
* The racial, gender and ethnic characteristics of the proposed subject population reflects the demographics of the University of Pittsburgh and the surrounding area and/or the patient population of the University of Pittsburgh Medical Center.
* The investigators shall attempt to recruit subjects in respective proportion to these demographics. No exclusion criteria shall be based on race, ethnicity, gender or HIV status.

Exclusion Criteria:

* Criteria for exclusion in the research study will be any pediatric patient, birth to 18 years, who are not in the active phase of craniofacial skeletal growth, and have not sustained a craniofacial fracture.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All races ages ranging from birth to 18 years who have sustained a craniofacial fracture.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
This protocol represents a descriptive and prospective, long-term, comprehensive growth and development study of the pediatric craniofacial skeleton following fracture | until subjects reach 18 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Losee, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospitla of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States